CLINICAL TRIAL: NCT01991990
Title: A Single Blind Phase IV Pharmacodynamic Study to Evaluate Neutrophil Distribution Kinetics and Function Following Single-Dose Tocilizumab Treatment in Healthy Subjects
Brief Title: A Pharmacodynamic Study to Evaluate Neutrophil Distribution Kinetics and Function Following Single-Dose RoActemra/Actemra (Tocilizumab) in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: WA29049
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Results first posted 2015-11-11 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- RoActemra/Actemra (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: placebo — Single i.v. infusion
  Arms: Placebo
Drug: tocilizumab [RoActemra/Actemra] — Single 8 mg/kg i.v. infusion
  Arms: RoActemra/Actemra

SUMMARY:
This Phase IV, single-blind , randomized, two-arm study will explore the pharmacodynamics effects of RoActemra/Actemra (tocilizumab) on neutrophil redistribution, function and survival in healthy subjects. Subjects will receive either a single dose of intravenous (IV) RoActemra/Actemra at a dose of 8 mg/kg over one hour on study Day 0 or placebo. Neutrophil kinetics data will be collected for all subjects up to Day 10 of the study. Following the last study visit on Day 10, all subjects will attend two further safety follow-up visits on Day 28 and Day 56.

ELIGIBILITY:
Inclusion Criteria:

* Male aged between 18 and 65 years inclusive
* Healthy as determined by screening assessments
* Body mass index (BMI) 18 to 30 kg/m2 inclusive
* Non-smoker
* Must agree to use a barrier method of contraception supplemented with spermicide during the treatment period and for at least 150 days after the last dose of study drug

Exclusion Criteria:

* Participation in a clinical study with an investigational drug within 3 months or at least 5 half-lives (whichever is longer) prior to dosing
* Current or past history of smoking within 6 months
* Previous exposure to therapeutic monoclonal antibodies in the past 6 months prior to screening
* Current or clinically significant history of any condition that, in the opinion of the investigator, would: place the subject at undue risk; invalidate the giving of informed consent; interfere with PK or PD data; or interfere with the ability of the subject to complete the study
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Any recurrent infections; infection requiring antibiotic treatment in the 6 weeks prior to dosing; mononucleosis in the 6 months prior to dosing; known HIV, Hepatitis B, or Hepatitis C; or active infection at the time of screening
* Active tuberculosis (TB) requiring treatment within the previous 3 years.
* Evidence of active malignant disease, malignancies diagnosed within the previous 10 years (except basal cell carcinoma of the skin that has been excised and cured), or breast cancer diagnosed within the previous 20 years
* Primary or secondary immunodeficiency
* Autoimmune disease
* Use or dependence on substance of abuse
* Alcohol abuse or average weekly intake greater than 2 units per day
* Screening or baseline resting heart rate < 45 or >90 beats per minute
* Major surgery within 8 weeks prior to screening
* Major illness in the 3 months prior to dosing
* Biliary obstruction
* Current or past history of diverticulitis

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Cambridge, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The screening visit was up to 3 weeks before randomization to the first dose of study medication. Out of 23 screened participants; 5 participants discontinued (4=met exclusion criteria; 1=withdrew), 18 participants were included.
Groups:
- Placebo: Participants received a single dose of placebo-matched to tocilizumab on Day 0.
- Tocilizumab: Participants received a single dose of intravenous (IV) tocilizumab (TCZ) at a dose of 8 milligrams (mg) per kilogram (kg) body weight infusion over 1 hour on Day 0.
Period: Overall Study
Arm/Group | Placebo | Tocilizumab
Started | 6 | 12
Completed | 6 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes all the randomized participants.
Groups:
- Tocilizumab: Participants received a single dose of IV TCZ at a dose of 8 mg/kg body weight infusion over 1 hour on Day 0.
- Total: Total of all reporting groups
Arm/Group | Placebo | Tocilizumab | Total
Number analyzed (Participants) | 6 | 12 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (11.0) | 34.5 (12.6) | 32.7 (12.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 12 | 18

OUTCOME MEASURES:

1. Primary Outcome: Neutrophil Redistribution Analysis on Day 4 (Neutrophil Nadir)
Description: On Day 4 participants had neutrophils isolated from 100 milliliters (mL) of acid-citrate dextrose (ACD)-anti-coagulated autologous venous blood and labeled in autologous plasma with up to 2.5 megaBecquerel (MBq) 111 Indium (111In)-tropolonate before being reinjected. Participants rested for 45 minutes (min) post-injection to allow for neutrophil equilibrium between the circulating and marginating neutrophil pools. Whole-body profiling was performed in a heavily shielded dedicated whole-body counter with 2 highly sensitive scintillation detectors with the recorded counts corrected for the physical decay of 111In to allow measurement of the effect of TCZ on the normal redistribution pattern of neutrophils and assessment of margination of neutrophils in the presence of TCZ. Distribution of radiolabelled neutrophils on Day 4 (45 min post re-injection) in the blood, liver/spleen and pelvic bone marrow, expressed as percentages of total body counts (TBCs).
Time Frame: Day 4
Population: Safety analysis population: Includes all the participants who received the single dose of randomized study medication. One participant in the polymorphonuclear leukocyte (PMN)-high group was excluded due to external contamination affecting profiling data.
Measure: Mean (Standard Error); unit: percentage of total body count
Groups:
- Tocilizumab (Polymorphonuclear Leukocyte (PMN)]-High Group): Participants who received a single dose of IV TCZ at a dose of 8 mg/kg body weight infusion over 1 hour on Day 0 and with less than or equal to (≤) 50% neutrophil count decrease at Day 4 relative to baseline were included in this group.
- Tocilizumab (PMN-Low Group): Participants who received a single dose of IV TCZ at a dose of 8 mg/kg body weight infusion over 1 hour on Day 0 and with greater than (>) 50% neutrophil count decrease at Day 4 relative to baseline were included in this group.
Arm/Group | Placebo | Tocilizumab (Polymorphonuclear Leukocyte (PMN)]-High Group) | Tocilizumab (PMN-Low Group)
Number analyzed (Participants) | 6 | 4 | 7
percentage of total body count
  Blood | 26.7 (4.7) | 26.5 (1.9) | 30.8 (5)
  Liver/Spleen | 50.4 (1.6) | 55 (3.1) | 52.4 (1.1)
  Pelvic marrow | 12.6 (0.9) | 11.7 (1) | 10.8 (1)

2. Primary Outcome: Neutrophil Redistribution Analysis on Day 5
Description: On Day 4 participants had neutrophils isolated from 100 mL of ACD-anti-coagulated autologous venous blood and labeled with up to 2.5 MBq 111In-tropolonate before being reinjected. Participants rested for 45 min post-injection to allow for neutrophil equilibrium between the circulating and marginating neutrophil pools. Whole-body profiling was performed in a heavily shielded dedicated whole-body counter with 2 highly sensitive scintillation detectors with the recorded counts corrected for the physical decay of 111In to allow measurement of the effect of TCZ on the normal redistribution pattern of neutrophils and assessment of margination of neutrophils in the presence of TCZ. Distribution of radiolabelled neutrophils and peak counts, on Day 5 (24-hours post re-injection) in liver/spleen and pelvic bone marrow were decay corrected and expressed as percentages of Day 4 (45 minutes post re-injection).
Time Frame: Day 5
Population: Safety analysis population. One participant in the PMN-high group was excluded due to external contamination affecting profiling data.
Measure: Mean (Standard Error); unit: percentage of Day 4 counts
Groups:
- Tocilizumab (PMN-High Group): Participants who received a single dose of IV TCZ at a dose of 8 mg/kg body weight infusion over 1 hour on Day 0 and ≤50% neutrophil count decrease at Day 4 relative to baseline were included in this group.
- Tocilizumab (PMN-Low Group): Participants who received a single dose of IV TCZ at a dose of 8 mg/kg body weight infusion over 1 hour on Day 0 and >50% neutrophil count decrease at Day 4 relative to baseline were included in this group.
Arm/Group | Placebo | Tocilizumab (PMN-High Group) | Tocilizumab (PMN-Low Group)
Number analyzed (Participants) | 6 | 4 | 7
percentage of Day 4 counts
  Liver/spleen peak counts (Day 5) | 91.0 (5.1) | 90.3 (5.0) | 105.2 (3.3)
  Pelvic peak counts (Day 5) | 187.8 (14.1) | 178.4 (18.9) | 129.1 (7.0)

3. Primary Outcome: Neutrophil Redistribution Analysis on Day 10
Description: On Day 4 participants had neutrophils isolated from 100 mL of ACD-anti-coagulated autologous venous blood and labeled with up to 2.5 MBq 111In-tropolonate before being reinjected. Participants rested for 45 min post-injection to allow for neutrophil equilibrium between the circulating and marginating neutrophil pools. Whole-body profiling was performed in a heavily shielded dedicated whole-body counter with 2 highly sensitive scintillation detectors with the recorded counts corrected for the physical decay of 111In to allow measurement of the effect of TCZ on the normal redistribution pattern of neutrophils and assessment of margination of neutrophils in the presence of TCZ. Distribution of radiolabelled neutrophils and peak counts, on Day 10 (6 days post re-injection) in liver/spleen and pelvic bone marrow were decay corrected and expressed as percentages of Day 4 (45 minutes post re-injection).
Time Frame: Day 10
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percentage of Day 4 counts
Groups:
- Tocilizumab (PMN-High Group): Participants who received a single dose of IV TCZ at a dose of 8 mg/kg body weight infusion over 1 hour on Day 0 and with ≤50% neutrophil count decrease at Day 4 relative to baseline were included in this group.
Arm/Group | Placebo | Tocilizumab (PMN-High Group) | Tocilizumab (PMN-Low Group)
Number analyzed (Participants) | 6 | 4 | 7
percentage of Day 4 counts
  Liver/spleen peak counts (Day 10) | 84.1 (6.2) | 76.6 (3.3) | 96.2 (2.9)
  Pelvic peak counts (Day 10) | 180.3 (12.9) | 175.6 (14.4) | 132.6 (5.0)

4. Primary Outcome: Neutrophil Phagocytosis: Change From Baseline to Nadir (Day 4) in the Percentage of eFluor670-Positive (eFluoro670+) Neutrophils
Description: Neutrophil phagocytosis was assessed by flow cytometry using heat-killed Staphylococcal pneumonia (S.pneumonia) bacteria labeled with eFluor670. Phagocytosis was quantified by measuring the eFluor670 fluorescence from neutrophils containing phagocytosed bacteria. Experiments were performed using neutrophils (PMN) only, PMN plus S. pneumonia at 4 degrees(˚) centigrade (C) (to control for non-specific bacterial adherence to PMN cell surface), and PMN plus S. pneumonia at 37˚C. Change from baseline in the percentage of eFluor670+ neutrophils was calculated on Day 4.
Time Frame: Baseline, Day 4
Population: Safety analysis population.
Measure: Mean (Standard Error); unit: percentage of eFlouro+ neutrophils
Arm/Group | Placebo | Tocilizumab (PMN-High Group) | Tocilizumab (PMN-Low Group)
Number analyzed (Participants) | 6 | 5 | 7
percentage of eFlouro+ neutrophils
  PMN only | 0 (0) | 0 (0) | 0 (0)
  PMN and S.pneumonia at 4˚C | -1 (1) | 2 (1) | 5 (2)
  PMN and S.pneumonia at 37˚C | 4 (2) | 7.5 (2) | 9 (2)

5. Primary Outcome: Neutrophil Phagocytosis: Change From Baseline to Nadir (Day 4) in Median Fluorescence Intensity (MFI) of eFluor670+ Neutrophils
Description: Neutrophil phagocytosis was assessed by flow cytometry using heat-killed Staphylococcal pneumonia bacteria labeled with eFluor670. Phagocytosis was quantified by measuring the eFluor670 fluorescence from neutrophils containing phagocytosed bacteria. Experiments were performed using neutrophils (PMN) only, PMN plus S. pneumonia at 4˚C (to control for non-specific bacterial adherence to PMN cell surface), and PMN plus S. pneumonia at 37˚C. Change from baseline in the eFluor670+ MFI was calculated on Day 4.
Time Frame: Baseline, Day 4
Population: Safety analysis population
Measure: Mean (Standard Error); unit: median fluoresence intensity
Arm/Group | Placebo | Tocilizumab (PMN-High Group) | Tocilizumab (PMN-Low Group)
Number analyzed (Participants) | 6 | 5 | 7
median fluoresence intensity
  PMN only | -1 (3) | 2 (7) | 2 (2)
  PMN and S.pneumonia at 4˚C | -2 (3) | 39 (18) | 32 (7)
  PMN and S.pneumonia at 37˚C | 685 (443) | 979 (350) | 810 (217)

6. Primary Outcome: Neutrophil Respiratory Burst: Change From Baseline to Nadir (Day 4) in the Production of Reactive Oxygen Species as Measured by Chemiluminescence (Relative Light Units - Absolute)
Description: Neutrophils generate a respiratory burst using reactive oxygen species (ROS) to kill invading pathogens. When luminol is used as a substrate for ROS, a chemical reaction is produced resulting in photon emission (chemiluminescence) in primed and unprimed neutrophils following formyl-methionyl-leucyl-phenylalanine (fMLP) stimulation which is quantifiable. fMLP stimulation of the respiratory burst is mediated through activation of nicotinamide adenine dinucleotide phosphate (NADPH) oxidase in primed neutrophils. The maximal fMLP response is observed in primed neutrophils and is an ex vivo measure of the capacity of neutrophils to respond to pathogenic stimuli. In the current experiments, neutrophils were primed with tumor necrosis factor alpha (TNFα). Light emission was recorded on a luminometer. Absolute change from baseline in the production of ROS on Day 4 was reported.
Time Frame: Baseline, Day 4
Population: Safety analysis population
Measure: Mean (Standard Error); unit: relative light units
Arm/Group | Placebo | Tocilizumab (PMN-High Group) | Tocilizumab (PMN-Low Group)
Number analyzed (Participants) | 6 | 5 | 7
relative light units
  Unprimed neutrophils | -16710 (12346) | -5553 (6409) | -2766 (3291)
  TNF α primed neutrophils | 82465 (16727) | -45257 (17540) | 64072 (16130)

7. Primary Outcome: Neutrophil Survival: Change From Baseline to the Nadir (Day 4) in the Percentage of Apoptotic Neutrophils as Measured by Microscopic Morphology
Description: Neutrophil apoptosis was measured using microscopy method with slides stained with Diff-Quik (modified Wright Giemsa stain) and morphology examined under oil immersion light microscopy with 100 times magnification. Neutrophils constitutively undergo apoptosis when cultured ex vivo, and this can be delayed by the addition of agents such as granulocyte-macrophage colony-stimulating factor (GM-CSF) or TNFα. Apoptotic neutrophils were characterized with dark and pyknotic nuclei compared to the viable neutrophils. Change from baseline in the percentage of apoptotic neutrophils on Day 4 measured by microscopy is reported.
Time Frame: Baseline, Day 4
Population: Safety analysis population
Measure: Mean (Standard Error); unit: percentage of apoptotic neutrophils
Arm/Group | Placebo | Tocilizumab (PMN-High Group) | Tocilizumab (PMN-Low Group)
Number analyzed (Participants) | 6 | 5 | 7
percentage of apoptotic neutrophils
  Untreated neutrophils | -6.0 (3.0) | -1.8 (4.0) | -6.0 (5.0)
  GM-CSF neutrophils | -1.0 (1.0) | -7.0 (5.0) | -12.0 (6.0)
  TNFα neutrophils | -2.0 (4.0) | 3.0 (4.0) | -4.0 (5.0)

8. Primary Outcome: Neutrophil Survival: Change From Baseline to the Nadir in the Percentage of Apoptotic Neutrophils as Measured by Flow Cytometry
Description: Ageing neutrophils translocate phosphatidylserine from the inner leaflet of the plasma membrane to the outer leaflet during the early stages of apoptosis. This translocation can be measured due to the affinity of Annexin V (AV) to bind exposed phosphatidylserine. Propidium Iodide (PI) is normally membrane-impermeable but enters cells in late apoptosis when their plasma membrane becomes leaky. Neutrophils constitutively undergo apoptosis when cultured ex vivo, and this can be delayed by the addition of agents such as granulocyte-macrophage colony-stimulating factor (GM-CSF) or TNFα. Apoptosis was assessed by flow cytometry with fluorescein isocyanate-labeled recombinant human AV (AV-FITC) and PI staining and the change from baseline in the percentage of apoptotic neutrophils on Day 4 measured by flow cytometry is reported.
Time Frame: Baseline, Day 4
Population: Safety analysis population
Measure: Mean (Standard Error); unit: percentage of apoptotic neutrophils
Arm/Group | Placebo | Tocilizumab (PMN-High Group) | Tocilizumab (PMN-Low Group)
Number analyzed (Participants) | 6 | 5 | 7
percentage of apoptotic neutrophils
  Untreated neutrophils | -5.0 (2.0) | -8.0 (4.0) | -7.0 (5.0)
  GM-CSF neutrophils | -4.0 (2.0) | -13.0 (4.0) | -9.0 (8.0)
  TNFα neutrophils | -3.0 (4.0) | 3.0 (2.0) | 3.0 (5.0)

9. Primary Outcome: Neutrophil Morphology: Change From Baseline to Nadir in the Number of Neutrophils With Shape Change Measured Using Flow Cytometry
Description: Neutrophil shape change is an indicator of the chemotactic ability of neutrophils to respond to and migrate to sites of inflammation. For determination of neutrophil shape change, fresh (0 min control), phosphate-buffered saline (PBS) control (30 min control) and formyl-methionyl-leucyl-phenylalanine (fMLP)-stimulated (30 min fMLP) PMNs (at 5 × 10^6 PMNs/ milliliter [mL]) were fixed with CellFIX (organic solvent used as fixative for adherent cells), 90 microliters (μL) transferred to each sample tube, and cold PBS added to stop further reaction. Shape change was assessed by measuring forward scatter (FSC) on flow cytometry. Change from baseline in the number of neutrophils with shape change on Day 4 was reported.
Time Frame: Baseline, Day 4
Population: Safety analysis population
Measure: Mean (Standard Error); unit: neutrophils with shape change
Arm/Group | Placebo | Tocilizumab (PMN-High Group) | Tocilizumab (PMN-Low Group)
Number analyzed (Participants) | 6 | 5 | 7
neutrophils with shape change
  0 min control | 1613 (842) | -359 (2613) | 4790 (1341)
  30 min control | 4882 (3069) | -2309 (4439) | 8814 (3016)
  30 min fMLP | -1889 (2800) | -1667 (4093) | 1524 (3515)

10. Primary Outcome: Neutrophil Morphology: Change From Baseline to the Nadir (Day 4) in the Percentage of Neutrophils With Shape Change Measured by Flow Cytometry (FSC-High Cells)
Description: Neutrophil shape change is an indicator of the chemotactic ability of neutrophils to respond to and migrate to sites of inflammation. For determination of neutrophil shape change, fresh (0 min control), PBS control (30 min control) and fMLP-stimulated (30 min fMLP) PMNs (at 5 × 10^6 PMNs/ mL) were fixed with CellFIX, 90 μL transferred to each sample tube, and cold PBS added to stop further reaction. Shape change was assessed by measuring FSC on flow cytometry. Change from baseline in the percentage of neutrophils with shape change on Day 4 was reported.
Time Frame: Baseline, Day 4
Population: Safety analysis population
Measure: Mean (Standard Error); unit: percentage of shape changed neutrophils
Arm/Group | Placebo | Tocilizumab (PMN-High Group) | Tocilizumab (PMN-Low Group)
Number analyzed (Participants) | 6 | 5 | 7
percentage of shape changed neutrophils
  0 min control | 14.0 (11.0) | 0.0 (3.0) | 2.0 (2.0)
  30 min control | 17.0 (8.0) | 1.0 (4.0) | 6.0 (3.0)
  30 min fMLP | 1.0 (3.0) | 0.0 (2.0) | -1.0 (3.0)

11. Primary Outcome: Neutrophil Morphology: Change From Baseline to the Nadir (Day 4) in the Percentage of Neutrophils With Shape Change Measured by Microscopic Morphology
Description: Neutrophil shape change is an indicator of the chemotactic ability of neutrophils to respond to and migrate to sites of inflammation. For determination of neutrophil shape change, fresh (0 min control), PBS control (30 min control) and fMLP-stimulated (30 min fMLP) PMNs (at 5 × 10^6 PMNs/ mL) were fixed with CellFIX, 90 μL transferred to each sample tube, and cold PBS added to stop further reaction. Shape change was assessed by microscopy with neutrophils classified as shape-changed if they contained > 1 cell surface bleb or irregularity and change from baseline in percentage of neutrophil with shape change on Day 4 was reported.
Time Frame: Baseline, Day 4
Population: Safety analysis population
Measure: Mean (Standard Error); unit: percentage of shape changed neutrophils
Arm/Group | Placebo | Tocilizumab (PMN-High Group) | Tocilizumab (PMN-Low Group)
Number analyzed (Participants) | 6 | 5 | 7
percentage of shape changed neutrophils
  0 min control | 12.0 (10.0) | -3.0 (4.0) | 0.0 (2.0)
  30 min control | 13.0 (11.0) | -2.0 (4.0) | -1.0 (1.0)
  30 min fMLP | 2.0 (6.0) | 4.0 (5.0) | -1.0 (3.0)

12. Primary Outcome: Absolute Median Fluorescence Intensities of Neutrophil Adhesion Molecules
Description: Neutrophil surface receptor expression may be used to characterize the activation status of neutrophils. Fresh (0 min), PBS control (30 min) and fMLP-stimulated (30 min) PMNs (5 × 10^6 PMNs/mL) were fixed with CellFIX, and 90 μL transferred to each tube containing antibody mixture (2 μL cluster of differentiation [CD] 11b-brilliant violet (BV) 421, 2 μL CD16-FITC, 5 μL CD62L-allophycocyanin (APC) and 5 μL CD162-phycoerythrin [PE]) or isotype control mixture of equivalent volumes. After 30 minutes of incubation on ice and in the dark, cold PBS was added to stop further reaction. Surface marker expressions were quantified by flow cytometry.
Time Frame: Day 4
Population: Safety analysis population
Measure: Mean (Standard Error); unit: median fluoresence intensity
Arm/Group | Placebo | Tocilizumab (PMN-High Group) | Tocilizumab (PMN-Low Group)
Number analyzed (Participants) | 6 | 5 | 7
median fluoresence intensity
  CD11b - 0 min control | 12633 (2062) | 15751 (2043) | 17764 (1910)
  CD11b - 30 min control | 13144 (2416) | 16047 (2058) | 18134 (1836)
  CD11b - 30 min fMLP | 39629 (2699) | 44481 (5049) | 41339 (2723)
  CD16 - 0 min control | 15822 (741) | 16872 (1874) | 15901 (1476)
  CD16 - 30 min control | 13771 (706) | 14885 (1744) | 13475 (1269)
  CD16 - 30 min fMLP | 17145 (884) | 18229 (2613) | 14707 (2205)
  CD62L - 0 min control | 563 (37) | 650 (201) | 767 (65)
  CD62L - 30 min control | 493 (38) | 588 (181) | 615 (37)
  CD62L - 30 min fMLP | 6 (3) | 5 (9) | 9 (12)
  CD162 - 0 min control | 3393 (454) | 3253 (895) | 3849 (314)
  CD162 - 30 min control | 3088 (433) | 2972 (820) | 3355 (347)
  CD162 - 30 min fMLP | 1571 (219) | 1568 (472) | 1733 (154)

ADVERSE EVENTS:
Time Frame: From baseline to 8 weeks of safety follow-up (approximately 8 months)
Arm/Group | Placebo | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 3/6 | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | Tocilizumab (N=12)
Aspartate aminotransferase increased (Investigations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Eosinophil count increased (Investigations) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.